CLINICAL TRIAL: NCT05301283
Title: Phase 2 Clinical Trial of Radiomic Habitat-Directed Radiation Dose Escalation for High-Grade Soft Tissue Sarcoma
Brief Title: Habitat Escalated Adaptive Therapy (HEAT), With Neoadjuvant Radiation for Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21136
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: High Grade Sarcoma
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants will receive pretreatment diagnostic MRIs to generate MRI habitats (images of tumor regions/subregions in different sequences). These images will identify radioresistant cells within the tumor to allow for more precise and higher doses of radiation to the resistant cells.
  Participants will then be treated with neoadjuvant external beam radiation by using the intensity modulated radiation (IMRT) technique, with dose painting (simultaneous integrated boost/SIB) to 70 Gray Units (Gy), 60 Gy, and 50 Gy in 25 fractions for habitats 1, 2, and 3, respectively.
  Interventions: Radiation: Intensity Modulated Radiation Therapy (IMRT); Diagnostic Test: MRI

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy (IMRT) — Participants will be treated with intensity modulated radiation therapy (IMRT) with photons, which is FDA (U.S. Food and Drug Administration) approved radiation delivery system.
Diagnostic Test: MRI — Participants will receive pretreatment diagnostic MRIs to generate MRI habitats. These images will identify radioresistant cells within tumor.

SUMMARY:
The purpose of the study is to utilize radiomic images to precisely locate areas of tumor that can be treated with dose escalation radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* For women of childbearing potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 52 weeks after the end of radiation.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner 52 weeks after radiation.
* Agreement to adhere to Lifestyle Considerations (as outlined in protocol) throughout study duration.
* Pathologically (histologically or cytologically) proven diagnosis of high-grade (grade 2 or 3) Soft Tissue Sarcoma (STS) of the deep trunk and/or extremity. Clinical evidence should be documented, and may consist of pathology or imaging, and should be sufficient to estimate the size of the primary (for T stage)
* Primary site deemed resectable prior to the start of trial
* American Joint Committee on Cancer (AJCC) 8th edition staging T1-4 N0 M0, no evidence of distant metastases
* Patients must have clinically or radiographically evident measurable disease at the primary site.
* Pre-Radiation Therapy (RT) MRI within 4 weeks of the start of RT.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 3.
* Deemed a surgical candidate
* Participant agrees to blood and plasma preservation for future analysis.

Exclusion Criteria:

* Contraindications to an MRI
* Positive urine pregnancy test
* Gross total excision of primary STS, including an unplanned excision
* Superficial sarcoma located primarily in the subcutaneous or cutaneous tissue
* Prior radiation to the region of the study cancer that would result in overlap of radiation therapy fields.
* Participants with a medical condition or social situation that, at the discretion of the principal investigator, would preclude them from completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Favorable Pathologic Response (FPR) | Week 10
  Percentage of participants with Favorable Pathologic Response (FPR): tumor necrosis >/= 95% at time of surgery. FPR is associated with improved R0 resection rates, local control, distant control, and overall survival. Therefore, FPR acts as an early surrogate for outcome.

SECONDARY OUTCOMES:
Percentage of tumor with clear margin and positive margin | Weeks 10-13
  Review of final tumor margin of the surgical specimen, defined as tumor at ink margin, will be conducted by pathologist. A clear margin (R0) or a positive margin (R1/R2) will be designated, along with the location of the margin, which will be radiographically correlated to the habitat . Surgical margins are independent predictors for local control.

OTHER OUTCOMES:
Disease Control Rate | Up to 6 months
  Disease control rate defined as the sum of complete response, partial response, and stable disease rates.
Overall Survival | Up to 8 months
  Overall Survival defined as the time from date of initial treatment to date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Arash O Naghavi, MD, MS, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naghavi AO, Bryant JM, Kim Y, Weygand J, Redler G, Sim AJ, Miller J, Coucoules K, Michael LT, Gloria WE, Yang G, Rosenberg SA, Ahmed K, Bui MM, Henderson-Jackson EB, Lee A, Lee CD, Gonzalez RJ, Feygelman V, Eschrich SA, Scott JG, Torres-Roca J, Latifi K, Parikh N, Costello J. Habitat escalated adaptive therapy (HEAT): a phase 2 trial utilizing radiomic habitat-directed and genomic-adjusted radiation dose (GARD) optimization for high-grade soft tissue sarcoma. BMC Cancer. 2024 Apr 9;24(1):437. doi: 10.1186/s12885-024-12151-7. PMID 38594603